CLINICAL TRIAL: NCT03130673
Title: Hip Fracture Epidemiology at Hospital Regional Rafael Hernandez. September 2014 to March 2015.
Brief Title: Challenges of Hip Fracture Care in Developing Countries. Experience at a Level 3 Center in Panama
Status: Completed | Type: Observational
Sponsor: Hospital del Niño "Dr. José Renán Esquivel" (Other)
Responsible Party: Principal Investigator, Arizt De Leon Robles, Orthopedic Resident, Hospital del Niño "Dr. José Renán Esquivel"
Other Study IDs: HRRH
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Hip Fractures
Keywords: hip fracture; trochanteric fracure; subtrocantheric fracture; femoral head fracture; epidemiology
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hip fracture: fracture of proximal femur

SUMMARY:
An observational study using the information records at the Hospital Regional Rafael Hernandez, in Chiriqui, Panama, that will help to analyze the epidemiology and early treatments results of hip fracture patients treated in this institution.

DETAILED DESCRIPTION:
Hip fractures are a major public health concern due to increasing ageing of the population, rising costs and associated morbidity and mortality. The problem is more serious in developing countries, because of limited economic and technical resources available. The aim of the following study is to analyze the epidemiology and early treatment results of hip fracture patients treated in our unit.

This study will be done at the Hospital Rafael Hernandez Regional Hospital, a third level facility located in the province of Chiriqui, Republic of Panama. It is a retrospective observational study.

For this the study will use the hospital records, including imaging studies were reviewed, including the Singh Index, and all relevant data will be analyzed with SPSS 21 software.

ELIGIBILITY:
Inclusion Criteria:

* All hip fractures

Exclusion Criteria:

* All other fractures and no recorded survey

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the Hip fractures in Hospital Regional Rafael Hernandez from september 2014 until march 2015
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Anatomical classified action of the Fracture | 6 months
  kind of proximal femoral fracture as sub trochanteric, intertrochanteric or subcapital

SECONDARY OUTCOMES:
Sex | 6 months
  male or female
Age | 6 months
  years old of the patient when he or she has the fracture
Comorbidities | 6 months
  Diseases of the patient (diabetes, hight blood pressure, others)
Energy of Trauma | 6 months
  IF it was high energy or low energy trauma
Average length of stay | 6 months
  Time frame that the patient stayed at the hospital
Osteoporosis | 6 months
  Severe, mild, light

CONTACTS AND LOCATIONS:
Overall Officials: Arizt De Leon, MD, Principal Investigator — orthopaedic surgeon
Locations (1):
- Panama Children Hospital, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ethgen O, Tellier V, Sedrine WB, De Maeseneer J, Gosset C, Reginster JY. Health-related quality of life and cost of ambulatory care in osteoporosis: how may such outcome measures be valuable information to health decision makers and payers? Bone. 2003 Jun;32(6):718-24. doi: 10.1016/s8756-3282(03)00089-9. PMID 12810180
- [Background] Clark, P.; Chico, G.; Carlos F y cols (2013) Osteoporosis En América Latina: Revisión De Panel De Expertos. Medwave. 13(8):E5791
- [Background] U.S. Census Bureau, (2011) International Data Base. Retrieved from http://www.census.gov/
- [Background] Nacionales DC, Szpila B, Ungaro R, Lopez MC, Zhang J, Gentile LF, Cuenca AL, Vanzant E, Mathias B, Jyot J, Westerveld D, Bihorac A, Joseph A, Mohr A, Duckworth LV, Moore FA, Baker HV, Leeuwenburgh C, Moldawer LL, Brakenridge S, Efron PA. A Detailed Characterization of the Dysfunctional Immunity and Abnormal Myelopoiesis Induced by Severe Shock and Trauma in the Aged. J Immunol. 2015 Sep 1;195(5):2396-407. doi: 10.4049/jimmunol.1500984. Epub 2015 Aug 5. PMID 26246141
- [Background] Bank, I. (1994). Latin America in Graphs: Demographic and Economic Trends 1972-1992. Population And Development Review, 20(3), 677. http://dx.doi.org/10.2307/2137618.
- [Background] Glenn, V. (2006). International Data Base (IDB) 2006, 188 International Data Base (IDB). URL: http://www.census.gov/ipc/www/idbnew.html: International Programs Center, US Census Bureau Last visited November 2005. Reference Reviews, 20(4), 19-19.
- [Background] Chue de Coto E. [The incidence of hip fractures in pre- and postmenopausal women in Panama]. Rev Med Panama. 1997 Jan;22(1):30-8. Spanish. PMID 9805092
- [Background] Chue de Coto E. [Osteopenia and osteoporosis in postmenopausal women in Panama]. Rev Med Panama. 2000;25:34-7. Spanish. PMID 15881746
- [Background] Moja L, Piatti A, Pecoraro V, Ricci C, Virgili G, Salanti G, Germagnoli L, Liberati A, Banfi G. Timing matters in hip fracture surgery: patients operated within 48 hours have better outcomes. A meta-analysis and meta-regression of over 190,000 patients. PLoS One. 2012;7(10):e46175. doi: 10.1371/journal.pone.0046175. Epub 2012 Oct 3. PMID 23056256
- [Background] Zanchetta J, Macdonald S. (2012) The Latin America Regional Audit. Epidemiology, Costs & Burden Of Osteoporosis In 2012. Switzerland: International Osteoporosis Foundation.
- [Background] Clark P, Carlos F, Vázquez-Martínez JL. (2010) Epidemiology, Costs And Burden Of Osteoporosis In Mexico. Arch Osteoporos. 5:9-17
- [Background] Sandoval, Ricardo. Epidemiologia y Costos de las Fracturas de Cadera en egresados del Complejo Hospitalario Metropolitano De La Caja De Seguro Social, Año 1990.
- [Background] Morales-Torres J, Gutierrez-Urena S; Osteoporosis Committee of Pan-American League of Associations for Rheumatology. The burden of osteoporosis in Latin America. Osteoporos Int. 2004 Aug;15(8):625-32. doi: 10.1007/s00198-004-1596-3. Epub 2004 Mar 20. PMID 15292978
- [Background] Etxebarria-Foronda I, Mar J, Arrospide A, Ruiz de Eguino J. [Cost and mortality associated to the surgical delay of patients with a hip fracture. Spain]. Rev Esp Salud Publica. 2013 Nov-Dec;87(6):639-49. doi: 10.4321/S1135-57272013000600008. Spanish. PMID 24549361
- [Background] von Friesendorff M, Besjakov J, Akesson K. Long-term survival and fracture risk after hip fracture: a 22-year follow-up in women. J Bone Miner Res. 2008 Nov;23(11):1832-41. doi: 10.1359/jbmr.080606. PMID 18597630
- [Background] Bartonicek J, Bartoska R. [Trochanteric fractures - anatomy and classification]. Rozhl Chir. 2013 Oct;92(10):581-8. Czech. PMID 24295482
- [Background] Ahmad T, Ashraf U, Irfan O, Muhammad ZA. Trends in management of neck of femur fracture. J Pak Med Assoc. 2015 Nov;65(11 Suppl 3):S163-5. PMID 26878511
- [Background] Dhanwal DK, Dennison EM, Harvey NC, Cooper C. Epidemiology of hip fracture: Worldwide geographic variation. Indian J Orthop. 2011 Jan;45(1):15-22. doi: 10.4103/0019-5413.73656. PMID 21221218
- [Background] Karampampa K, Andersson T, Drefahl S, Ahlbom A, Modig K. Does improved survival lead to a more fragile population: time trends in second and third hospital admissions among men and women above the age of 60 in Sweden. PLoS One. 2014 Jun 9;9(6):e99034. doi: 10.1371/journal.pone.0099034. eCollection 2014. PMID 24911650
- [Background] Singh M, Nagrath AR, Maini PS. Changes in trabecular pattern of the upper end of the femur as an index of osteoporosis. J Bone Joint Surg Am. 1970 Apr;52(3):457-67. No abstract available. PMID 5425640
- [Background] Pahor M, Guralnik JM, Ambrosius WT, Blair S, Bonds DE, Church TS, Espeland MA, Fielding RA, Gill TM, Groessl EJ, King AC, Kritchevsky SB, Manini TM, McDermott MM, Miller ME, Newman AB, Rejeski WJ, Sink KM, Williamson JD; LIFE study investigators. Effect of structured physical activity on prevention of major mobility disability in older adults: the LIFE study randomized clinical trial. JAMA. 2014 Jun 18;311(23):2387-96. doi: 10.1001/jama.2014.5616. PMID 24866862
- [Background] Martínez López, R., Moreno Navarro, J., Goide Linares, E., & Fernández García, D. (2012). Caracterización Clinico epidemiológica de pacientes con Fracturas de Cadera. Medisan, 16(2), 182-188.
- [Background] Muñoz,S., Lavanderos, J.,& Vilches, L. (2008). Fractura de Cadera. Cuad Cir (Valdivia), 22(1), 73-81.
- [Background] Becarra-Rojas F, Jupari M (2011) Epidemiology of Osteoporosis In Perú. Bone 29:294-313
- [Background] Sicras-Mainar A, Navarro-Artieda R, Ibanez-Nolla J. [Use of resources and costs associated to fractures in Spanish women]. Rev Peru Med Exp Salud Publica. 2012 Jul-Sep;29(3):350-6. doi: 10.1590/s1726-46342012000300009. Spanish. PMID 23085796
- [Background] Riera-Espinoza G. Epidemiology of osteoporosis in Latin America 2008. Salud Publica Mex. 2009;51 Suppl 1:S52-5. doi: 10.1590/s0036-36342009000700009. PMID 19287895
- [Background] Orces CH. Epidemiology of hip fractures in Ecuador. Rev Panam Salud Publica. 2009 May;25(5):438-42. doi: 10.1590/s1020-49892009000500009. PMID 19695134
- [Background] Vanzant EL, Hilton RE, Lopez CM, Zhang J, Ungaro RF, Gentile LF, Szpila BE, Maier RV, Cuschieri J, Bihorac A, Leeuwenburgh C, Moore FA, Baker HV, Moldawer LL, Brakenridge SC, Efron PA; Inflammation and Host Response to Injury Investigators. Advanced age is associated with worsened outcomes and a unique genomic response in severely injured patients with hemorrhagic shock. Crit Care. 2015 Mar 4;19(1):77. doi: 10.1186/s13054-015-0788-x. PMID 25880307
- [Background] Berggren M, Stenvall M, Englund U, Olofsson B, Gustafson Y. Co-morbidities, complications and causes of death among people with femoral neck fracture - a three-year follow-up study. BMC Geriatr. 2016 Jun 3;16:120. doi: 10.1186/s12877-016-0291-5. PMID 27260196
- [Background] Ercolano, M. A., Drnovsek, M. L., & Gauna, A. (2012). Fractura de Cadera en los Hospitales Públicos de la Argentina. Revista Argentina de Endocrinología y Metabolismo, 49(1), 3-11.
- [Background] Méndez-Lavergne O, Medina M, Avid J. (2011) Perfil de Pacientes con Fractura de Cadera. Hospital El Vigía. Eneroa-Agosto 2011. Rev MédCient; 24(2):3-11.
- [Background] Tortosa, Eric. (2004) Epidemiología de las Fracturas de Cadera en el Hospital Regional Rafael Hernández. Estudio Prospectivo, Junio 2003 - Marzo 2004.
- [Background] Etxebarria-Foronda I, Caeiro-Rey JR, Larrainzar-Garijo R, Vaquero-Cervino E, Roca-Ruiz L, Mesa-Ramos M, Merino Perez J, Carpintero-Benitez P, Fernandez Cebrian A, Gil-Garay E. [SECOT-GEIOS guidelines in osteoporosis and fragility fracture. An update]. Rev Esp Cir Ortop Traumatol. 2015 Nov-Dec;59(6):373-93. doi: 10.1016/j.recot.2015.05.007. Epub 2015 Jul 29. No abstract available. Spanish. PMID 26233814
- [Background] Jiménez C, Camacho D, Sepúlveda M. (2013) Aproximación epidemiológica de las fracturas de cadera en Chile. Rev Chil Ortop Traumatol 54 (3): 126-30.
- [Background] Carriero FP, Christmas C. In the clinic. Hip fracture. Ann Intern Med. 2011 Dec 6;155(11):ITC6-1-ITC6-15; quiz ITC6-16. doi: 10.7326/0003-4819-155-11-201112060-01006. No abstract available. PMID 22147729
- [Background] Chang KP, Center JR, Nguyen TV, Eisman JA. Incidence of hip and other osteoporotic fractures in elderly men and women: Dubbo Osteoporosis Epidemiology Study. J Bone Miner Res. 2004 Apr;19(4):532-6. doi: 10.1359/JBMR.040109. Epub 2004 Jan 5. PMID 15005838
- [Background] Khan SK, Shirley MD, Glennie C, Fearon PV, Deehan DJ. Achieving best practice tariff may not reflect improved survival after hip fracture treatment. Clin Interv Aging. 2014 Dec 1;9:2097-102. doi: 10.2147/CIA.S65736. eCollection 2014. PMID 25489240
- [Background] Simunovic N, Devereaux PJ, Bhandari M. Surgery for hip fractures: Does surgical delay affect outcomes? Indian J Orthop. 2011 Jan;45(1):27-32. doi: 10.4103/0019-5413.73660. PMID 21221220
- [Background] Nazrun AS, Tzar MN, Mokhtar SA, Mohamed IN. A systematic review of the outcomes of osteoporotic fracture patients after hospital discharge: morbidity, subsequent fractures, and mortality. Ther Clin Risk Manag. 2014 Nov 18;10:937-48. doi: 10.2147/TCRM.S72456. eCollection 2014. PMID 25429224
- [Background] Amigo P, Rodríguez M. (2012) Complicaciones intrahospitalarias de los pacientes intervenidos de fractura de cadera. Rev Med Electron 30(5):e1.
- [Background] Dinamarca-Montecinos JL, Amestica-Lazcano G, Rubio-Herrera R, Carrasco-Buvinic A, Vasquez A. [Hip fracture. Experience in 647 Chilean patients aged 60 years or more]. Rev Med Chil. 2015 Dec;143(12):1552-9. doi: 10.4067/S0034-98872015001200008. Spanish. PMID 26928617
- [Background] PALOMINO, Lourdes; RAMIREZ, Rubén; VEJARANO, Julio y TICSE, Ray. (2016) Fractura de cadera en el adulto mayor: la epidemia ignorada en el Perú. Acta méd. peruana , vol.33, n.1, pp. 15-20 .
- [Background] Azagra R, Roca G, Encabo G, Prieto D, Aguye A, Zwart M, Guell S, Puchol N, Gene E, Casado E, Sancho P, Sola S, Toran P, Iglesias M, Sabate V, Lopez-Exposito F, Ortiz S, Fernandez Y, Diez-Perez A. Prediction of absolute risk of fragility fracture at 10 years in a Spanish population: validation of the WHO FRAX tool in Spain. BMC Musculoskelet Disord. 2011 Jan 28;12:30. doi: 10.1186/1471-2474-12-30. PMID 21272372
- [Background] Pedrera-Zamorano JD, Lavado-Garcia JM, Moran JM. Comment on Sanfelix-Genoves et al.: Prevalence of osteoporotic fracture risk factors and antiosteoporotic treatments in the Valencia region, Spain. The baseline characteristics of the ESOSVAL cohort. Osteoporos Int. 2013 Jun;24(6):1923-4. doi: 10.1007/s00198-012-2145-0. Epub 2012 Sep 29. No abstract available. PMID 23052931
- [Result] Kanis JA, Oden A, McCloskey EV, Johansson H, Wahl DA, Cooper C; IOF Working Group on Epidemiology and Quality of Life. A systematic review of hip fracture incidence and probability of fracture worldwide. Osteoporos Int. 2012 Sep;23(9):2239-56. doi: 10.1007/s00198-012-1964-3. Epub 2012 Mar 15. PMID 22419370